CLINICAL TRIAL: NCT02250690
Title: Transcranial Direct Current Stimulation (tDCS) Associated With Gait Training in Improving Motor Function in Parkinson's Disease
Brief Title: Neuromodulation on Motor Function in Parkinson's Disease
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Adriana Carla Costa Ribeiro Clementino, Transcranial direct current stimulation (tDCS) associated with gait training in improving motor function in Parkinson's disease., Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Parkinson_tDCS_Gait_Impairment
Record Dates: First submitted 2014-03-31; First posted 2014-09-26 (Estimated); Last update posted 2014-09-26 (Estimated); Status verified 2014-07

CONDITIONS: Idiopathic Parkinsons Disease
Keywords: idiopathic PD; Hoehn and Yahr stage I to III; stable medication usage; age 40 to 80 years; absence of cognitive impairment
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- experimental group - tDCS (Experimental): The tDCS intervention occur at 10 sessions of intervention where electrodes are connected to head specifically in supplementary motor area placed at 2 cm in front of vertex. The clinical stimulator (NeuroConn, Germany) provided the direct current using two silicon-sponge electrodes with a surface area of 35 cm2 (5 × 7cm) embedded in a saline-soaked solution. Immediately after 13 minutes of tDCS application, patient was submitted to gait training three times a week during 4 weeks with visuals cues. The patients were asked to walk along at a 7 meters rubber carpet to at different speed, forward and backward gait, side walk during thirty minutes with three intervals of two minutes. The patient may be at on state of drug administration and the training is applied by another physiotherapist.
  Interventions: Device: experimental group - tDCS
- Control group (tDCS sham) (Sham Comparator): The sham character is ensured by the stimulation time, once the device is programmed to turn off 30 seconds after the beginning of stimulation. The current is switched in ascending ramp mode for 10 seconds until 2 mili ampere and a descending ramp similar also for 10 seconds will be used until the end of stimulation. The sham stimulation is commonly perceived by the patient as the actual treatment and all procedures for the application of the technique should be similar to those adopted for the active stimulation. Immediately after tDCS stimulation, the gait training consisting of a protocol based on sensory cues for 30 minutes is administered three times a week for four weeks. Sham stimulation will be held for 30 seconds in order to mimic the perceived lowering effect of ramp current.
  Interventions: Device: Control group (tDCS sham)

INTERVENTIONS:
Device: experimental group - tDCS
  Arms: experimental group - tDCS
Device: Control group (tDCS sham)
  Arms: Control group (tDCS sham)

SUMMARY:
The aims of the present study was to analyze the effect of consecutive sessions of Transcranial direct current stimulation associated to kinesiotherapy about gait performance of Parkinson' s disease. For this, the primary outcome was evaluation of gait performance by means of space and temporal parameters as speed (meter/second ), stride frequency (steps/min) and stride length (m). The secondary outcome is motor cortex excitability which is analyzed by means of single pulse transcranial magnetic stimulation (TMS) intends to determine: motor evoked potential amplitude (MEP) and rest motor threshold (rMT).

DETAILED DESCRIPTION:
This study consist by interventions involving screening followed by evaluation, where volunteers were subjected to the many tests: history, session III of the Unified Scale Modified Parkinson's Disease - Unified Parkinson 's Disease Rating Scale, Ten meters walk test - Walk Test 10 meters and shoot gait, (using Studio Version 8 software). On the same day, the subjects underwent assessment of brain excitability to determine motor threshold and amplitude of the motor evoked potential (MEP). The randomization of the volunteers was conducted by an external search through opaque envelopes ordered according to a random distribution. The subjects were divided into two groups : control group , this group submitted to Transcranial Stimulation sessions a sham Continuous Current (sham tDCS) and gait training , and Experimental group, subjected to the stimulation by Transcranial Direct Current sessions (active tDCS ) and gait training.

ELIGIBILITY:
Inclusion Criteria:

* Main eligibility criteria were idiopathic Parkinson's disease
* Both sex
* Hoehn and Yahr stage I to III
* Showing mild to severe gait disturbances
* Stable medication usage
* Age 40 to 80 years
* And absence of cognitive impairment and disorders interfering with participation in cueing therapy.

Exclusion Criteria:

* Presence of chronic disabling pathologies of lower limb
* Presence of pacemaker or severe cardiovascular conditions
* A history of tumor, prior neurosurgical brain
* Intervention, or severe cardiovascular conditions, including the presence of a pacemaker
* A diagnosis of epilepsy or major psychiatric disorders.
* Participants with other neurological, muscular, or psychiatric disorders (e.g. peripheral neuropathies, uncorrected visual problems, hearing problems, vestibular dysfunction, stroke, seizure, migraine, or frequent severe headaches) were excluded.
* Participants with surgical implants, significant postural tremor, dyskinesia, severe freezing or dementia were also excluded.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2013-09; Primary Completion 2014-10 (Estimated); Study Completion 2014-11 (Estimated)

PRIMARY OUTCOMES:
Change on Bradykinesia | This outcome will be measure before and after each session, before ten sessions, 1 and 2 months after ten session
  This outcome will be measure in three different moments of evaluation and at all interventions (sessions) days - before and after intervention. Beyond these evaluations, the voluntairs will be evaluate at: T1- before ten sessions; T2- Immediately after ten sessions and T3- after a period of 1 month without intervention.

SECONDARY OUTCOMES:
Change on Cortical excitability | The evaluation occur in 3 different moments: before and after each session, after a period of 1 month without intervention. This outcome will be measure at all intervention and evaluation days
  The secondary outcome measures will be done using amplitude of Motor Evoked Potential (MEP) and rest Motor Threshold (rMT) elicited by transcranial magnetic stimulation (TMS) by means of Neuro-MS device of Neurosoft.

OTHER OUTCOMES:
Change on Balance | This outcome will be measure before ten sessions, 1 and 2 months after ten session
  Berg Balance scale (BBS) is measured asking to the patient for change posture in sit position for search balance during transferences and standing with one foot at single or double support, with open and closed eyes, narrow support base body, rotation around the own body axis; take up an object at floor and others. This outcome is done using a scale with scores range from 0 to 56.